CLINICAL TRIAL: NCT03699891
Title: Evaluation of the Fortilink IBF System With TETRAfuse Technology
Acronym: ENTRUST
Status: Completed | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1103
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Cervical and Lumbar Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fortilink IBF System with TETRAfuse Technology — Cervical and lumbar fusion

SUMMARY:
This is a multi-center, post-market, retrospective study to collect safety and performance data for patients implanted with the Fortilink IBF System.

DETAILED DESCRIPTION:
This is a multi-center, post-market, retrospective study to collect safety and performance data for patients implanted with the Fortilink IBF System.

The study will include up to 110 patients at up to 8 US sites. All patients implanted with the Fortilink System at a site will be included in the data collection. The goal is to collect data for at least 100 subjects, but the sample size will be capped at 110 to ensure that all patients at a given site are included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have had an attempted implant of the Fortilink IBF System

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient must have had an attempted implant of the Fortilink IBF System
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Safety outcomes associated with use of the Fortlink System | Up to 1 year
  Safety assessment includes evaluation of all adverse events or complications related to the procedure and post-operative adverse events.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles Orthopedic Institute, Sherman Oaks, California
  - Rocky Mountain Spine, Lone Tree, Colorado
  - Florida Back Institute, Boca Raton, Florida
  - Spine Institute of South Florida, Delray Beach, Florida
  - OrthoBethesda, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No